CLINICAL TRIAL: NCT05593419
Title: Selecting Patients Who May Benefit From Immunotherapy by Tissue-based Biomarkers
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, Shen Lin, Professor, Peking University
Other Study IDs: CGOG-GMAP 1.0
Record Dates: First submitted 2022-10-21; First posted 2022-10-25 (Actual); Last update posted 2022-10-25 (Actual); Status verified 2022-10

CONDITIONS: Gastric Cancer Patients Received Immunotherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Immunotherapy Group
  Interventions: Device: TIIC signature

INTERVENTIONS:
Device: TIIC signature — Collect tumor tissue of 300 gastric cancer patients at treatment baseline, samples will be transferred to central lab to detect the density and spatial proximity of certain immune cells infiltrated in tumor by multi complex immunohistochemistry, and evaluate patients' TIIC signature.Tumor response evaluation will be performed after two cycles of therapy by CT/MRI based on RECIST.Clinical data, including tumor stage,metastaticorgan ,regimen, objective response, progression free survival, overall survival, etc, will be collected according to study protocol.

SUMMARY:
We have established a machine learning model based on effective TIIC signature which could select GC patients who may benefit from immunotherapy.

The current study aims to enroll 300 GC patients as a validation cohort to vertify the accuracy of TIIC signature in predicting immunotherapy efficacy

ELIGIBILITY:
Inclusion Criteria:

* Having signed informed consent
* Age:18-80 years old
* Histologically confirmed gastric adenocarcinoma
* Unresectable recurrent or metastatic gastric cancer
* Previous neo-adjuvant or adjuvant treatment for gastric cancer, if applicable, more than 6 months
* Measurable disease according to the RECIST criteria
* Karnofsky performance status ≥70
* Life expectancy of ≥3 month
* No prior radiotherapy except radiotherapy at non-target lesion of the study more than 4 weeks
* ALT and AST<2.5 times ULN (≤5 times ULN in patients with liver metastases)
* Serum albumin level ≥3.0g/dL
* Serum AKP < 2.5 times ULN
* Serum creatinine <ULN, and CCr < 60ml/min
* Bilirubin level < 1.5 ULN
* WBC>3,000/mm3, absolute neutrophil count ≥2000/mm3, platelet>100,000/mm3, Hb>9g/dl

Exclusion Criteria:

* Previous systemic therapy for metastatic gastric cancer
* Surgery (excluding diagnostic biopsy) within 4 weeks prior to study entry Contraindications of nuclear magnetic resonance image such as fitment of cardiac pacemaker , nerve stimulator, or aneurysm clip, and metallic foreign body in eye ball and so on.
* Allergic constitution or allergic history to protium biologic product or any investigating agents.
* Severe heart disease or such history as recorded congestive heart failure, uncontrolled cardiac arrhythmia, angina pectoris needing medication, cardiac valve disease, severe abnormal ECG findings, cardiac infarction , or retractable hypertension.
* Pregnancy or lactation period
* Other previous malignancy within 5 year, except non-melanoma skin cancer
* Legal incapacity

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients in this study were enrolled by the Department of gastrointestinal oncology, Peking University Cancer Hospital & Institute for conventional therapy or clinical trials
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2022-10-31 (Estimated); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
TIIC signature | Treatment baseline
  Density and spatial proximity of 4 kinds of immune cells involved in TIIC signature infiltrate in tumor at treatment baseline will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Cancer Hospital, Beijing, China